CLINICAL TRIAL: NCT05086978
Title: Novel Clinical Utility of Retinal Imaging in Patients With Heart Failure: A Pilot Study
Brief Title: Novel Clinical Utility of Retinal Imaging in Patients With Heart Failure
Status: Enrolling by invitation | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Wilson Tang, Principal Investigator, The Cleveland Clinic
Other Study IDs: 21-940
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Heart Failure
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart Failure out-patients: Subjects with heart failure of any etiology
- Heart Failure in-patients: Subjects with heart failure of any etiology

SUMMARY:
Endothelial dysfunction and microvascular disease have been shown to play an important role in both the development and progression of heart failure. Retinal imaging provides a unique opportunity to non-invasively assess retinal microcirculation. Leveraging the non-invasiveness and relative ease of use of retinal imaging, we propose to investigate its clinical utility in assessing endothelial/microvascular dysfunction across the spectrum of heart failure. We aim to test the hypothesis that the degree of abnormality in retinal vessels is associated with heart failure disease severity, endothelial/microvascular dysfunction, and, potentially, treatment responses.

DETAILED DESCRIPTION:
This is a human study to test the hypothesis that the degree of abnormality in retinal vessels is associated with heart failure disease severity, endothelial/microvascular dysfunction, and, potentially, treatment responses. Previous epidemiology studies have shown an association between ophthalmic measurements like retinal vessel caliber, retinal microvascular signs, and retinopathy diagnosed from conventional digitized retinal imaging, and the risk of heart failure, as well as alterations in left ventricular structure and function, and even altered filling pressure. Automatic detection software for retinal vessel caliber measurement is widely available, and deep learning algorithms have already enabled reliable detection of retinopathy from captured retinal images. Optical Coherence Tomography (OCT) is an imaging technology that allows for noninvasive, non-contact, high-resolution, cross-sectional imaging of tissue in real time (1). OCT angiography is a new development in OCT imaging that provides visualization of microvascular flow in the retinae of human eyes without the need for intravenous injection of a contrast dye. Several OCT angiography (OCTA) methods allow for three-dimensional noninvasive microvascular visualization. The Zeiss® VisuScout 100, used in the pilot phase of the study, is a handheld retinal camera, commercially available and is already in clinical use at the Cleveland Clinic by Cole Eye Institute specialists for bedside consultations. However, the use of retinal imaging in risk stratifying cardiovascular diseases is unknown, in large part because routine capturing of these images at the point of care is not performed. Novel applications of this non-invasive screening strategy beyond routine ophthalmology-based evaluation may pave the way to scalable population health screening or disease monitoring initiatives. We have established laboratory procedures and equipment for all proposed biomarker evaluations and have published work supporting their mechanistic link to pathophysiologic processes.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or above; have been diagnosed with HF of any etiology or healthy control; able to provide informed consent and comply with study protocol; able to undergo retinal evaluation using a handheld, automated, non-mydriatric retinal camera; and able to provide written informed consent.

Exclusion Criteria:

* pregnancy or planned pregnancy; photosensitive epilepsy; significant ophthalmologic conditions such as cataract, glaucoma, blindness, or progressive diabetic retinopathy; having undergone retinal laser photocoagulation; any condition which, in the judgment of the investigator, would place a patient at undue risk by being enrolled in the trial, or cause inability to comply with the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Heart Failure subjects (any etiology)
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2022-02-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2027-01-01 (Estimated)

PRIMARY OUTCOMES:
Retinal measurements and heart failure severity | 4 years
  To generate the methodologies and establish workflow, and to generate preliminary data to demonstrate the association of retinal measurements with heart failure disease severity.
Retinal measurements and exercise capacity | 4 years
  To generate the methodologies and establish workflow, and to generate preliminary data to demonstrate the association of retinal measurements with exercise capacity represented by 6 Minute Walk Test distance

SECONDARY OUTCOMES:
Blood analysis | 4 years
  Blood samples may be collected to assess for asymmetric dimethylarginine levels (ADMA, a surrogate of endothelial dysfunction)
Urine analysis | 4 years
  Urine samples may be collected to obtain urine albumin/creatinine ratio (UACR) for microalbuminuria (a surrogate of microvascular disease)

CONTACTS AND LOCATIONS:
Overall Officials: W. H. Wilson Tang, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Marti CN, Gheorghiade M, Kalogeropoulos AP, Georgiopoulou VV, Quyyumi AA, Butler J. Endothelial dysfunction, arterial stiffness, and heart failure. J Am Coll Cardiol. 2012 Oct 16;60(16):1455-69. doi: 10.1016/j.jacc.2011.11.082. Epub 2012 Sep 19. PMID 22999723
- [Background] Goto I, Katsuki S, Ikui H, Kimoto K, Mimatsu T. Pathological studies on the intracerebral and retinal arteries in cerebrovascular and noncerebrovascular diseases. Stroke. 1975 May-Jun;6(3):263-9. doi: 10.1161/01.str.6.3.263. PMID 50653
- [Background] Tanaka M, Fujiwara H, Onodera T, Wu DJ, Matsuda M, Hamashima Y, Kawai C. Quantitative analysis of narrowings of intramyocardial small arteries in normal hearts, hypertensive hearts, and hearts with hypertrophic cardiomyopathy. Circulation. 1987 Jun;75(6):1130-9. doi: 10.1161/01.cir.75.6.1130. PMID 3552306
- [Background] Wong TY, Rosamond W, Chang PP, Couper DJ, Sharrett AR, Hubbard LD, Folsom AR, Klein R. Retinopathy and risk of congestive heart failure. JAMA. 2005 Jan 5;293(1):63-9. doi: 10.1001/jama.293.1.63. PMID 15632337
- [Background] Cheung N, Bluemke DA, Klein R, Sharrett AR, Islam FM, Cotch MF, Klein BE, Criqui MH, Wong TY. Retinal arteriolar narrowing and left ventricular remodeling: the multi-ethnic study of atherosclerosis. J Am Coll Cardiol. 2007 Jul 3;50(1):48-55. doi: 10.1016/j.jacc.2007.03.029. Epub 2007 Jun 18. PMID 17601545
- [Background] Chandra A, Seidelmann SB, Claggett BL, Klein BE, Klein R, Shah AM, Solomon SD. The association of retinal vessel calibres with heart failure and long-term alterations in cardiac structure and function: the Atherosclerosis Risk in Communities (ARIC) Study. Eur J Heart Fail. 2019 Oct;21(10):1207-1215. doi: 10.1002/ejhf.1564. Epub 2019 Aug 1. PMID 31373139
- [Background] Chung YR, Park SJ, Moon KY, Choi SA, Lim HS, Park SW, Kim JH, Lee K. Diabetic retinopathy is associated with diastolic dysfunction in type 2 diabetic patients with non-ischemic dilated cardiomyopathy. Cardiovasc Diabetol. 2017 Jul 6;16(1):82. doi: 10.1186/s12933-017-0566-y. PMID 28683825